CLINICAL TRIAL: NCT02133365
Title: Atrial Fibrillation, Cardiac Symptoms, and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Meghan Kolodziej, Associate Psychiatrist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000363
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Anxiety
MeSH Terms: conditions — Atrial Fibrillation; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness and Interoceptive Exposure (Active Comparator): Atrial fibrillation patients will receive 4-5 manualized, individualized sessions of Mindfulness and Interoceptive Exposure.
  Interventions: Behavioral: Mindfulness and Interoceptive Exposure
- Medical care as usual (No Intervention): Atrial fibrillation patients will receive medical and cardiac care as usual.

INTERVENTIONS:
Behavioral: Mindfulness and Interoceptive Exposure — The Mindfulness and Interoceptive Exposure intervention will be delivered in 4-5 manualized, individualized therapy sessions, of 1.5 hours - 2 hours each. The intervention is comprised of four established cognitive-behavioral strategies: psychoeducation, mindfulness, interoceptive exposure and skills generalization.
  Arms: Mindfulness and Interoceptive Exposure

SUMMARY:
This is an investigation of a mindfulness and interoceptive exposure intervention in patients with atrial fibrillation, to decrease anxiety sensitivity, symptom burden, and atrial fibrillation recurrence.

DETAILED DESCRIPTION:
Patients with atrial fibrillation (AF) have a poorer quality of life and have elevated rates of anxiety. Higher anxiety and somatization has been associated with more severe AF symptoms. Increased anxiety symptoms have also been associated with increased medical visits for AF management. Some studies show that anxiety may increase the risk of AF recurrence following medical intervention, including increasing AF recurrence after circumferential pulmonary vein ablation. Growing evidence suggests a pressing need to treat anxiety and improve quality of life among AF patients, yet few data exist about how to accomplish this. Mindfulness-based behavioral treatments offer promise in this regard.

Interoceptive Exposure (IE) is an evidence-based cognitive behavioral intervention to address intolerance of anxiety-related physical sensations, commonly seen in panic disorder and other anxiety disorders. It involves systematically and repeatedly inducing feared physical sensations to promote increased tolerance and reduced distress associated with these symptoms.

Mindfulness is defined as paying attention to the present moment in an open and nonjudgmental way. Mindfulness-based behavioral interventions have been successfully applied in various psychiatric and medical patient populations, including cardiac patients. Two meta-analyses suggest that mindfulness-based interventions are moderately effective for reducing distress related to physical or psychosomatic illnesses.

The investigators of this study hypothesize that a mindfulness and IE intervention will decrease anxiety, AF symptoms and AF recurrence, and will improve quality of life among patients with AF.

This is a pilot, prospective trial of a mindfulness and IE intervention in patients with AF. The mindfulness and IE intervention will be delivered in four to five, manualized, individual sessions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients
* At least 18 years of age
* Clinical diagnosis of Atrial Fibrillation
* Literacy and fluency in English
* Ability to return to the hospital for study visits
* Score ≥ 24 on the Anxiety Sensitivity Index-3.

Exclusion Criteria:

* Medical co-morbidity sufficient to confound the outcome variables
* Medical co-morbidity for which the experimental treatment is contraindicated
* Clinically significant cognitive impairment
* Known unavailability for follow-up in the ensuing 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-09; Primary Completion 2017-03 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Cardiac symptoms as measured by the Cardiac Symptom Questionnaire (CSQ). | 3 months
  The CSQ is a 15 item, self-report, symptom inventory with responses scored on a Likert scale

SECONDARY OUTCOMES:
Cardiac anxiety as measured by the Cardiac Anxiety Questionnaire (CAQ-R) | 3 months
Anxiety sensitivity as measured by the Anxiety Sensitivity Index-3 (ASI-3) | 3 months
Health related quality of life as measured by the Atrial Fibrillation Effect on Quality of Life (AFEQT) | 3 months
Atrial fibrillation severity | 3 months
  Atrial fibrillation severity as measured by routine clinical ambulatory monitoring with event recorders and other routine electrocardiographic monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan S Kolodziej, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Van Gelder IC, Hagens VE, Bosker HA, Kingma JH, Kamp O, Kingma T, Said SA, Darmanata JI, Timmermans AJ, Tijssen JG, Crijns HJ; Rate Control versus Electrical Cardioversion for Persistent Atrial Fibrillation Study Group. A comparison of rate control and rhythm control in patients with recurrent persistent atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1834-40. doi: 10.1056/NEJMoa021375. PMID 12466507
- [Background] Hagens VE, Vermeulen KM, TenVergert EM, Van Veldhuisen DJ, Bosker HA, Kamp O, Kingma JH, Tijssen JG, Crijns HJ, Van Gelder IC; RACE study group. Rate control is more cost-effective than rhythm control for patients with persistent atrial fibrillation--results from the RAte Control versus Electrical cardioversion (RACE) study. Eur Heart J. 2004 Sep;25(17):1542-9. doi: 10.1016/j.ehj.2004.06.020. PMID 15342174
- [Background] Gehi AK, Sears S, Goli N, Walker TJ, Chung E, Schwartz J, Wood KA, Guise K, Mounsey JP. Psychopathology and symptoms of atrial fibrillation: implications for therapy. J Cardiovasc Electrophysiol. 2012 May;23(5):473-8. doi: 10.1111/j.1540-8167.2011.02264.x. Epub 2012 Mar 19. PMID 22429764
- [Background] Yu SB, Hu W, Zhao QY, Qin M, Huang H, Cui HY, Huang CX. Effect of anxiety and depression on the recurrence of persistent atrial fibrillation after circumferential pulmonary vein ablation. Chin Med J (Engl). 2012 Dec;125(24):4368-72. PMID 23253703
- [Background] Craske MG, Barlow DH. (2007). Mastery of your anxiety and panic: Therapist guide (2nd Ed). New York, NY: Oxford University Press
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Kabat-Zinn J. (1990) Full catastrophe living: Using the wisdom of your body and mind to face stress, pain and illness. New York: Delacourt.
- [Background] Nyklicek I, Dijksman SC, Lenders PJ, Fonteijn WA, Koolen JJ. A brief mindfulness based intervention for increase in emotional well-being and quality of life in percutaneous coronary intervention (PCI) patients: the MindfulHeart randomized controlled trial. J Behav Med. 2014 Feb;37(1):135-44. doi: 10.1007/s10865-012-9475-4. Epub 2012 Nov 23. PMID 23180285
- [Background] Carlson LE, Ursuliak Z, Goodey E, Angen M, Speca M. The effects of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients: 6-month follow-up. Support Care Cancer. 2001 Mar;9(2):112-23. doi: 10.1007/s005200000206. PMID 11305069
- [Background] Roth B, Robbins D. Mindfulness-based stress reduction and health-related quality of life: findings from a bilingual inner-city patient population. Psychosom Med. 2004 Jan-Feb;66(1):113-23. doi: 10.1097/01.psy.0000097337.00754.09. PMID 14747645
- [Background] Speca M, Carlson LE, Goodey E, Angen M. A randomized, wait-list controlled clinical trial: the effect of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients. Psychosom Med. 2000 Sep-Oct;62(5):613-22. doi: 10.1097/00006842-200009000-00004. PMID 11020090
- [Background] Ledesma D, Kumano H. Mindfulness-based stress reduction and cancer: a meta-analysis. Psychooncology. 2009 Jun;18(6):571-9. doi: 10.1002/pon.1400. PMID 19023879
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Nyklicek I, Kuijpers KF. Effects of mindfulness-based stress reduction intervention on psychological well-being and quality of life: is increased mindfulness indeed the mechanism? Ann Behav Med. 2008 Jun;35(3):331-40. doi: 10.1007/s12160-008-9030-2. Epub 2008 Jun 6. PMID 18535870
- [Background] Grossman P, Niemann L, Schmidt S, Walach H. Mindfulness-based stress reduction and health benefits. A meta-analysis. J Psychosom Res. 2004 Jul;57(1):35-43. doi: 10.1016/S0022-3999(03)00573-7. PMID 15256293